CLINICAL TRIAL: NCT00733525
Title: Stepped Care vs Best Available Care for Bulimia Nervosa
Brief Title: Effectiveness of Stepped Care Versus Best Available Care for Bulimia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9802M00108; R01MH059304 (NIH); R01MH059303 (NIH); R01MH059301 (NIH); R01MH059100 (NIH); DSIR 83-ATAS (Other Grant/Funding Number: Foundation)
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Eating Disorders
Keywords: Bulimia Nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia Nervosa | interventions — Cognitive Behavioral Therapy; Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stepped Care (Experimental): Participants will receive guided self-help with nine clinician checkups, followed by fluoxetine if nonresponsive, followed by cognitive behavioral therapy if still nonresponsive.
  Interventions: Behavioral: Cognitive Behavioral Therapy; Drug: Fluoxetine; Behavioral: Guided Self-Help
- Cognitive Behavioral Therapy (Active Comparator): Participants will receive 20 sessions of cognitive behavioral therapy with the addition of fluoxetine at interim points.
  Interventions: Behavioral: Cognitive Behavioral Therapy; Drug: Fluoxetine

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Therapy focusing on skills needed to alter eating patterns
Drug: Fluoxetine — 20 mg/day of fluoxetine, which can be incrementally increased to 80 mg/day
  Other Names: Prozac
Behavioral: Guided Self-Help — Manual designed to impart teachings of cognitive behavioral therapy
  Arms: Stepped Care

SUMMARY:
This study will compare the medical and cost effectiveness of a stepped approach, including self-help and drug therapies, to the current best available care for bulimia nervosa.

DETAILED DESCRIPTION:
The eating disorder bulimia nervosa (BN) is estimated to exist in 1 % to 2 % of women from the ages of 15 to 30, and bulimic behaviors occur in many more who do not develop the disorder. Characteristic symptoms include binge eating and self-induced vomiting. Research indicates that cognitive behavioral therapy (CBT), paired with use of the antidepressant fluoxetine, is the treatment of choice for BN. However, a survey of doctoral level psychologists dealing with eating disorders found that 78% of clinicians had no training in CBT for eating disorders, with 72% also untrained in the alternative, interpersonal therapy. Self-help manuals based on CBT have been developed as a treatment option for those without access to a clinician trained in CBT for eating disorders. Studies of these manuals suggest that self-guided therapy is as effective as CBT for some individuals. Additionally, although little research has examined cost effectiveness for treatment of eating disorders, a self-help approach may be more cost effective than CBT. This study will test whether self-help therapy, in the context of a stepped treatment plan involving check-ins with a clinician and possible drug treatment, can be an effective alternative, medically and economically, to traditional CBT.

Participants at four treatment sites will be screened for diagnosis, health, and presence of other conditions through assessments in standardized questionnaires, clinical interviews, and a blood test. Participants who pass the screening will be randomly assigned to one of two treatment sequences. In the first sequence, participants will be given twenty 50-minute sessions of individual CBT treatment over 18 weeks, focusing on altering eating behaviors. If participants do not have an adequate initial response to treatment by session six, they will be offered a trial of fluoxetine in addition to their continued CBT treatment. If they do not meet response criteria at the end of the 18 weeks of CBT treatment, they will again be given the option of taking or continuing to take fluoxetine until the termination of the study. The second sequence will begin with a specially designed self-help program aimed at teaching the same skills that will be taught in CBT sessions. Participants will have nine 30-minute checkup sessions with a therapist over 18 weeks. Participants who do not respond adequately to the treatment after 10 weeks will be given the option of taking fluoxetine. Participants without sufficient recovery at the end of 18 weeks will be given the option of undergoing the first treatment sequence.

Assessments of costs and health will be made at five points: the beginning of the study, and at the study visits on Week 10, Week 18, Week 36, and Week 62. Multiple assessments will be used to test health, including eating disorder symptoms, presence of other psychopathology and personality factors, social and interpersonal functioning, and quality of life. Eating disorder symptoms will be evaluated through clinical interview, questionnaires, and weight fluctuations. Treatment variables will also be assessed, with particular interest in the measure of patient knowledge of CBT techniques, to determine how much information from the self-help manual is used and absorbed. For the cost benefit analysis, assessments will include cost of health care visits, medications, treatments, and time lost due to illness. Data on cost will be collected at study visits, except for time lost, which will be measured through a questionnaire completed by a family member once at baseline and once after 18 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bulimia nervosa

Exclusion Criteria:

* Weight less than 85% of ideal
* Current substance abuse or dependence
* Pregnant
* Currently receiving psychotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2000-09; Primary Completion 2005-04 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Eating disorders examination | Measured at baseline and Weeks 10, 18, 36, and 62

SECONDARY OUTCOMES:
Records of health care, medications, and treatments | Measured at baseline and Weeks 10, 18, 36, and 62
Height, weight, and body mass index | Measured at baseline, Week 8, and Week 62
Battery of self-report questionnaires | Measured at baseline and Weeks 10, 18, 36, and 62
Questionnaire on time lost to bulimia, completed by a family member | Measured at baseline and after 18 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Agras, MD, Study Chair — Stanford University
Locations (4):
- United States (4):
  - Stanford University, Palo Alto, California
  - University of Minnesota Minneapolis, MN, Minneapolis, Minnesota
  - Cornell University; White Plains, NY, White Plains, New York
  - University of North Dakota / Neuropsychiatric Research Institute, Fargo, North Dakota

REFERENCES:
- [Derived] Mitchell JE, Agras S, Crow S, Halmi K, Fairburn CG, Bryson S, Kraemer H. Stepped care and cognitive-behavioural therapy for bulimia nervosa: randomised trial. Br J Psychiatry. 2011 May;198(5):391-7. doi: 10.1192/bjp.bp.110.082172. Epub 2011 Mar 17. PMID 21415046